CLINICAL TRIAL: NCT05194033
Title: Efficacy and Safety of Oral Lactobacillus Plantarum GUANKE (CGMCC NO.21720) in Enhancement of Antibody Level After SARS-CoV-2 Vaccination: A Prospective, Randomized, Double-blind, Placebo-Controlled Trial (Trial 1)
Brief Title: Efficacy and Safety of Oral Lactobacillus Plantarum GUANKE (CGMCC NO.21720) in Enhancement of Antibody Level After SARS-CoV-2 Vaccination (Trial 1)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); Beijing Pinggu District Hospital (Other); Peking University Health Science Center Hospital (Unknown)
Responsible Party: Principal Investigator, Yangfeng Wu, Professor of Epidemiology and Sciences in Clincial Research, Peking University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: GUANKE-Trial 1
Record Dates: First submitted 2022-01-12; First posted 2022-01-18 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: SARS-CoV-2
Keywords: Probiotic; lactobacillus plantarum

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, double-blind, placebo parallel controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is double-blinded, which neither participants nor investigators know the results of intervention. In addition, laboratory test of blood samples will also be conducted without knowing the randomization results of participants to ensure the evaluation of outcome measure is objective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): The intervention group consumes oral probiotics 1 time/day for 7 consecutive days.
  Interventions: Dietary Supplement: Probiotics daily
- Placebos (Placebo Comparator): The placebo group consumes oral placebo 1 time/day for 7 consecutive days.
  Interventions: Dietary Supplement: Placebo daily

INTERVENTIONS:
Dietary Supplement: Probiotics daily — Probiotics 1 time/day for 7 consecutive days
  Arms: Probiotics
Dietary Supplement: Placebo daily — Placebo 1 time/day for 7 consecutive days
  Arms: Placebos

SUMMARY:
Preliminarily explore the effect of oral probiotics in SARS-CoV-2 serum neutralizing antibody titer level and T cell response level (spot formation cell counting).

Provide a reference for determining the appropriate oral regimen. Provide necessary parameters for estimating the sample size of confirmatory clinical trial.

DETAILED DESCRIPTION:
In selected communities or assigned clinical trial institutions, participants who had completed two doses of SARS-CoV-2 vaccination will be invited in this study. Informed consent form will give to potential participants with well explained of trial contents during baseline. Participants who gave their signed informed consent form will be blocked randomized in a 1:1 ratio to intervention group or placebo control group.

ELIGIBILITY:
Inclusion Criteria:

1. 18 ≤age ≤59 years;
2. Vaccinated with two doses of SARS-CoV-2 vaccine (manufactured by Sino Biopharmaceutical Limited or SINOVAC BIOTECH CO., LTD.) (≥6 months from the time of vaccination).
3. Not vaccinated third dose vaccination;
4. Voluntarily participate in the study with signed informed consent form.

Exclusion criteria:

1. Pregnancy or lactation period;
2. Infected with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV);
3. Plan to vaccinate third dose of SARS-CoV-2 vaccine within 2 months;
4. History of autoimmune diseases (e.g. rheumatoid arthritis, systemic lupus erythematosus, dry syndrome, etc.);
5. Previously infected with SARS-CoV-2 or close contact of SARS-CoV-2 infected individual;
6. Other SARS-CoV-2 vaccination history (not manufactured by Sino Biopharmaceutical Limited or SINOVAC BIOTECH CO., LTD.);
7. End-stage cancer or other terminal diseases with life expectancy <6 month;
8. History of severe cardiovascular and cerebrovascular diseases, such as heart failure, uncontrolled coronary heart disease, cardiomyopathy, uncontrolled arrhythmia,or history of myocardial or cerebral infarction within past six months;
9. Participating in other clinical trials.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-03-09 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
The serum neutralizing antibody level of SARS-CoV-2. | 8 weeks
  The serum neutralizing antibody level of SARS-CoV-2 is determined by serum neutralization test, which is used to determine the serum dilution that protects 50% cells from cytopathic effect.
T-cell response level | 8 weeks
  Test of T-cell response level by spot-forming cell(SFC) counting, using Champspot III enzyme-linked spot automated image analysis system.

SECONDARY OUTCOMES:
Antibody concentration | 8 weeks
  The binding antibody concentration of S protein IgG and IgA in SARS-CoV-2 serum.
PBMC transcriptome expression | 8 weeks
  The expression of PBMC transcriptome
Serum cytokines | 8 weeks
  The test of serum cytokines
Serum neutralizing antibody positive rate | 8 weeks
  The positive rate of serum neutralizing antibody.
Serum neutralizing antibody positive conversion rate | 8 weeks
  The positive conversion rate of serum neutralizing antibody.
Intestinal flora | 8 weeks
  The level of intestinal flora.
Fecal viable culture | 8 weeks
  The culture of fecal viable
Fecal specific binding antibody IgA | 8 weeks
  The specific binding antibody IgA of fecal
Blood pressure | 8 weeks
  The level of blood pressure.
Blood glucose | 8 weeks
  The level of blood glucose.
Blood lipid | 8 weeks
  The level of blood lipid.

OTHER OUTCOMES:
Safety indicators | 8 weeks
  Adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Yangfeng Wu, Principal Investigator — Peking University
Locations (2):
- China (2):
  - Beijing Pinggu Hospital, Beijing
  - Peking University Health Science Center Hospital, Beijing

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shrotri M, Navaratnam AMD, Nguyen V, Byrne T, Geismar C, Fragaszy E, Beale S, Fong WLE, Patel P, Kovar J, Hayward AC, Aldridge RW; Virus Watch Collaborative. Spike-antibody waning after second dose of BNT162b2 or ChAdOx1. Lancet. 2021 Jul 31;398(10298):385-387. doi: 10.1016/S0140-6736(21)01642-1. Epub 2021 Jul 17. No abstract available. PMID 34274038
- [Background] Naaber P, Tserel L, Kangro K, Sepp E, Jurjenson V, Adamson A, Haljasmagi L, Rumm AP, Maruste R, Karner J, Gerhold JM, Planken A, Ustav M, Kisand K, Peterson P. Dynamics of antibody response to BNT162b2 vaccine after six months: a longitudinal prospective study. Lancet Reg Health Eur. 2021 Nov;10:100208. doi: 10.1016/j.lanepe.2021.100208. Epub 2021 Sep 6. PMID 34514454
- [Background] Liu YW, Liong MT, Tsai YC. New perspectives of Lactobacillus plantarum as a probiotic: The gut-heart-brain axis. J Microbiol. 2018 Sep;56(9):601-613. doi: 10.1007/s12275-018-8079-2. Epub 2018 Aug 23. PMID 30141154
- [Background] Gorska A, Przystupski D, Niemczura MJ, Kulbacka J. Probiotic Bacteria: A Promising Tool in Cancer Prevention and Therapy. Curr Microbiol. 2019 Aug;76(8):939-949. doi: 10.1007/s00284-019-01679-8. Epub 2019 Apr 4. PMID 30949803
- [Background] Huang Y, Wang X, Wang J, Wu F, Sui Y, Yang L, Wang Z. Lactobacillus plantarum strains as potential probiotic cultures with cholesterol-lowering activity. J Dairy Sci. 2013 May;96(5):2746-53. doi: 10.3168/jds.2012-6123. Epub 2013 Mar 15. PMID 23498020
- [Background] Li J, Zhao F, Wang Y, Chen J, Tao J, Tian G, Wu S, Liu W, Cui Q, Geng B, Zhang W, Weldon R, Auguste K, Yang L, Liu X, Chen L, Yang X, Zhu B, Cai J. Gut microbiota dysbiosis contributes to the development of hypertension. Microbiome. 2017 Feb 1;5(1):14. doi: 10.1186/s40168-016-0222-x. PMID 28143587
- [Background] Palmu J, Salosensaari A, Havulinna AS, Cheng S, Inouye M, Jain M, Salido RA, Sanders K, Brennan C, Humphrey GC, Sanders JG, Vartiainen E, Laatikainen T, Jousilahti P, Salomaa V, Knight R, Lahti L, Niiranen TJ. Association Between the Gut Microbiota and Blood Pressure in a Population Cohort of 6953 Individuals. J Am Heart Assoc. 2020 Aug 4;9(15):e016641. doi: 10.1161/JAHA.120.016641. Epub 2020 Jul 21. PMID 32691653
- [Background] Khalesi S, Sun J, Buys N, Jayasinghe R. Effect of probiotics on blood pressure: a systematic review and meta-analysis of randomized, controlled trials. Hypertension. 2014 Oct;64(4):897-903. doi: 10.1161/HYPERTENSIONAHA.114.03469. Epub 2014 Jul 21. PMID 25047574
- [Background] Wu Y, Zhang Q, Ren Y, Ruan Z. Effect of probiotic Lactobacillus on lipid profile: A systematic review and meta-analysis of randomized, controlled trials. PLoS One. 2017 Jun 8;12(6):e0178868. doi: 10.1371/journal.pone.0178868. eCollection 2017. PMID 28594860
- [Background] Bock PM, Telo GH, Ramalho R, Sbaraini M, Leivas G, Martins AF, Schaan BD. The effect of probiotics, prebiotics or synbiotics on metabolic outcomes in individuals with diabetes: a systematic review and meta-analysis. Diabetologia. 2021 Jan;64(1):26-41. doi: 10.1007/s00125-020-05295-1. Epub 2020 Oct 13. PMID 33047170
- [Background] Seddik HA, Bendali F, Gancel F, Fliss I, Spano G, Drider D. Lactobacillus plantarum and Its Probiotic and Food Potentialities. Probiotics Antimicrob Proteins. 2017 Jun;9(2):111-122. doi: 10.1007/s12602-017-9264-z. PMID 28271469
- [Background] Kujawa-Szewieczek A, Adamczak M, Kwiecien K, Dudzicz S, Gazda M, Wiecek A. The Effect of Lactobacillus plantarum 299v on the Incidence of Clostridium difficile Infection in High Risk Patients Treated with Antibiotics. Nutrients. 2015 Dec 4;7(12):10179-88. doi: 10.3390/nu7125526. PMID 26690209
- [Background] Ducrotte P, Sawant P, Jayanthi V. Clinical trial: Lactobacillus plantarum 299v (DSM 9843) improves symptoms of irritable bowel syndrome. World J Gastroenterol. 2012 Aug 14;18(30):4012-8. doi: 10.3748/wjg.v18.i30.4012. PMID 22912552
- [Background] Fuentes MC, Lajo T, Carrion JM, Cune J. Cholesterol-lowering efficacy of Lactobacillus plantarum CECT 7527, 7528 and 7529 in hypercholesterolaemic adults. Br J Nutr. 2013 May 28;109(10):1866-72. doi: 10.1017/S000711451200373X. Epub 2012 Sep 28. PMID 23017585
- [Background] Miele E, Pascarella F, Giannetti E, Quaglietta L, Baldassano RN, Staiano A. Effect of a probiotic preparation (VSL#3) on induction and maintenance of remission in children with ulcerative colitis. Am J Gastroenterol. 2009 Feb;104(2):437-43. doi: 10.1038/ajg.2008.118. Epub 2009 Jan 20. PMID 19174792
- [Background] Szymanski H, Armanska M, Kowalska-Duplaga K, Szajewska H. Bifidobacterium longum PL03, Lactobacillus rhamnosus KL53A, and Lactobacillus plantarum PL02 in the prevention of antibiotic-associated diarrhea in children: a randomized controlled pilot trial. Digestion. 2008;78(1):13-7. doi: 10.1159/000151300. Epub 2008 Aug 14. PMID 18701826
- [Background] Liu YW, Liong MT, Chung YE, Huang HY, Peng WS, Cheng YF, Lin YS, Wu YY, Tsai YC. Effects of Lactobacillus plantarum PS128 on Children with Autism Spectrum Disorder in Taiwan: A Randomized, Double-Blind, Placebo-Controlled Trial. Nutrients. 2019 Apr 11;11(4):820. doi: 10.3390/nu11040820. PMID 30979038
- [Background] Hwang YH, Park S, Paik JW, Chae SW, Kim DH, Jeong DG, Ha E, Kim M, Hong G, Park SH, Jung SJ, Lee SM, Na KH, Kim J, Chung YC. Efficacy and Safety of Lactobacillus Plantarum C29-Fermented Soybean (DW2009) in Individuals with Mild Cognitive Impairment: A 12-Week, Multi-Center, Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Nutrients. 2019 Feb 1;11(2):305. doi: 10.3390/nu11020305. PMID 30717153
- [Background] Hakansson A, Andren Aronsson C, Brundin C, Oscarsson E, Molin G, Agardh D. Effects of Lactobacillus plantarum and Lactobacillus paracasei on the Peripheral Immune Response in Children with Celiac Disease Autoimmunity: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Nutrients. 2019 Aug 16;11(8):1925. doi: 10.3390/nu11081925. PMID 31426299
- [Background] Chong HX, Yusoff NAA, Hor YY, Lew LC, Jaafar MH, Choi SB, Yusoff MSB, Wahid N, Abdullah MFIL, Zakaria N, Ong KL, Park YH, Liong MT. Lactobacillus plantarum DR7 alleviates stress and anxiety in adults: a randomised, double-blind, placebo-controlled study. Benef Microbes. 2019 Apr 19;10(4):355-373. doi: 10.3920/BM2018.0135. Epub 2019 Mar 18. PMID 30882244
- [Background] Lee A, Lee YJ, Yoo HJ, Kim M, Chang Y, Lee DS, Lee JH. Consumption of Dairy Yogurt Containing Lactobacillus paracasei ssp. paracasei, Bifidobacterium animalis ssp. lactis and Heat-Treated Lactobacillus plantarum Improves Immune Function Including Natural Killer Cell Activity. Nutrients. 2017 May 31;9(6):558. doi: 10.3390/nu9060558. PMID 28561762
- [Background] Lew LC, Hor YY, Yusoff NAA, Choi SB, Yusoff MSB, Roslan NS, Ahmad A, Mohammad JAM, Abdullah MFIL, Zakaria N, Wahid N, Sun Z, Kwok LY, Zhang H, Liong MT. Probiotic Lactobacillus plantarum P8 alleviated stress and anxiety while enhancing memory and cognition in stressed adults: A randomised, double-blind, placebo-controlled study. Clin Nutr. 2019 Oct;38(5):2053-2064. doi: 10.1016/j.clnu.2018.09.010. Epub 2018 Sep 19. PMID 30266270
- [Background] Nam B, Kim SA, Park SD, Kim HJ, Kim JS, Bae CH, Kim JY, Nam W, Lee JL, Sim JH. Regulatory effects of Lactobacillus plantarum HY7714 on skin health by improving intestinal condition. PLoS One. 2020 Apr 10;15(4):e0231268. doi: 10.1371/journal.pone.0231268. eCollection 2020. PMID 32275691
- [Background] Kageyama Y, Nishizaki Y, Aida K, Yayama K, Ebisui T, Akiyama T, Nakamura T. Lactobacillus plantarum induces innate cytokine responses that potentially provide a protective benefit against COVID-19: A single-arm, double-blind, prospective trial combined with an in vitro cytokine response assay. Exp Ther Med. 2022 Jan;23(1):20. doi: 10.3892/etm.2021.10942. Epub 2021 Nov 2. PMID 34815772
- [Background] Lee MC, Tu YT, Lee CC, Tsai SC, Hsu HY, Tsai TY, Liu TH, Young SL, Lin JS, Huang CC. Lactobacillus plantarum TWK10 Improves Muscle Mass and Functional Performance in Frail Older Adults: A Randomized, Double-Blind Clinical Trial. Microorganisms. 2021 Jul 8;9(7):1466. doi: 10.3390/microorganisms9071466. PMID 34361902